CLINICAL TRIAL: NCT05415475
Title: A Safety and Efficacy Clinical Study of CEA-targeted CAR-T Therapy for CEA-positive Advanced Malignant Solid Tumors
Brief Title: Clinical Study of CEA-targeted CAR-T Therapy for CEA-positive Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC034
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Stomach Cancer; Pancreatic Cancer; Metastatic Tumor; Recurrent Cancer
Keywords: CAR-T; CEA; CEA-positive advanced malignant solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-10x107 copy/kg
  Interventions: Biological: CEA CAR-T cells
- intraperitoneal injection of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-10x107 copy/kg
  Interventions: Biological: CEA CAR-T cells

INTERVENTIONS:
Biological: CEA CAR-T cells — Administration method: intravenous infusion or intraperitoneal injection； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This trial is an open-label, single-arm clinical study. The main purpose is to verify the safety and efficacy of CAR-T cell preparations in the treatment of CEA-positive advanced malignant tumors, and to obtain the recommended dose and infusion scheme of CAR-T cell preparations for the treatment of patients with CEA-positive advanced malignant tumors.

DETAILED DESCRIPTION:
Carcinoembryonic antigen (CEA) is a classic tumor marker, which is positively expressed in a variety of digestive tract tumors. In normal tissue cells, only a small amount of CEA is expressed in the cell membrane of digestive tract cells. In the early clinical trials of CAR-T targeting CEA carried out by the technical partner, it was found that CAR-T cell preparations have a certain killing effect on CEA-positive tumor cells. At the same time, no serious CAR-T-related adverse events were found through dose-escalating infusion. In this study, through the optimization of the CAR structure and the improvement of the culture method, the killing ability and survival ability of the CAR-T cell preparation on tumor cells in vitro and in vivo were improved to further verify the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Advanced, metastatic or recurrent malignant tumors diagnosed by histology or pathology, mainly colorectal cancer, esophageal cancer, gastric cancer, and pancreatic cancer;
3. After receiving at least second-line standard treatment and failing (disease progression or intolerance, such as surgery, chemotherapy, radiotherapy, etc.) or lack of effective treatment methods;
4. Immunohistochemical staining of tumor samples within 3 months confirmed that the tumor was CEA positive (clear membrane staining, positive rate ≥ 10%); the patient's serum CEA should exceed 10ug/L.
5. At least one assessable lesion according to RECIST 1.1 criteria;
6. ECOG score 0-2 points;
7. No serious mental disorder;
8. Unless otherwise specified, the function of the vital organs of the subject shall meet the following conditions:

   1. Blood routine: white blood cells>2.0×109/L, neutrophils>0.8×109/L, lymphocytes cells>0.5×109/L, platelets>50×109/L, hemoglobin>90g/L;
   2. Cardiac function: echocardiography showed cardiac ejection fraction ≥50%, and no obvious abnormality was found on electrocardiogram;
   3. Renal function: serum creatinine≤2.0×ULN;
   4. Liver function: ALT and AST ≤3.0×ULN (for those with liver tumor infiltration, it can be relaxed to≤5.0×ULN);
   5. Total bilirubin≤2.0×ULN;
   6. Oxygen saturation > 92% in non-oxygen state.
9. Have apheresis or venous blood collection standards, and have no other contraindications for cell collection;
10. Subjects agree to use reliable and effective contraceptive methods for contraception within 1 year after signing the informed consent form to receiving CAR-T cell infusion (excluding rhythm contraception);
11. The patients themselves or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.

Exclusion Criteria:

1. Previous CAR-T therapy or other gene-modified cell therapy；
2. CNS metastases or meningeal metastases with clinical symptoms at the time of screening, or there is other evidence that the patient's central nervous system metastases or meningeal metastases have not been controlled, and are judged by the investigator to be unsuitable for inclusion;
3. Participated in other clinical studies within 1 month before screening;
4. vaccinated with live attenuated vaccine within 4 weeks before screening;
5. Received the following anti-tumor treatments before screening: Received chemotherapy, targeted therapy or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter);
6. Active infection or uncontrollable infection requiring systemic treatment;
7. Patients with intestinal obstruction, active gastrointestinal bleeding, or a history of gastrointestinal bleeding within 3 months;
8. Except for alopecia or peripheral neuropathy, the toxicity of previous anti-tumor therapy has not improved to the baseline level or ≤ grade 1;
9. Suffering from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment;
   3. Clinically significant ventricular arrhythmia, or history of syncope of unknown origin (caused by vasovagal except those caused by neurosis or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
10. Patients with active autoimmune disease, or other patients requiring long-term immunosuppressive therapy;
11. Suffering from other uncured malignant tumors in the past 3 years or at the same time, except cervical carcinoma in situ and basal cell carcinoma of the skin;
12. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer is greater than the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Virus (HCV) RNA test is greater than the normal range; human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
13. Women who are pregnant or breastfeeding;
14. Other investigators deem it unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CEA-CAR-T cells infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of CEA-CAR-T cells[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Disease control rate of CAR-T cell preparations in CEA-positive advanced malignancies [Effectiveness] | 3 months
  Disease control rate: including CR, PR and SD
Changes in serum tumor markers of CAR-T cell preparations in CEA-positive advanced malignancies [Effectiveness] | 3 months
  Changes in serum tumor markers：CEA、 CA199、 CA125
AUCS of CEA-CAR-T cells [Cell dynamics] | 1 years
  AUCS is defined as the area under the curve in 28 days and 90 days
CMAX of CEA-CAR-T cells [Cell dynamics] | 1 years
  CMAX is defined as the highest concentration of CEA-CAR-T cells expanded in peripheral blood
TMAX of CEA-CAR-T cells[Cell dynamics] | 1 years
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CEA-CAR-T cells[Cell dynamics] | 1 years
  The content of free CEA in peripheral blood at each time point measured by Chemiluminescence immunoassay

OTHER OUTCOMES:
Objective response rate (ORR) of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  Objective response rate includes：CR、PR
Duration of Response (DOR) of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression.
Overall survival(OS)of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 1 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause
Proportion of tumor cells in tumor tissue of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 years
  The rate of tumor cell in tumor tissue will be measured by biopsy and immunohistochemistry
CEA expression level of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 years
  The CEA expression in tumor tissue will be measured by biopsy and immunohistochemis
Changes in the number of tumor-infiltrating immune cells of CEA- CAR-T treatment in patients with CEA-positive | 1 years
  the number of tumor-infiltrating immune cells will be measured by biopsy and immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Jingwang Bi, M.D, Principal Investigator — Shandong Second Provincial General Hospital
Locations (1):
- Shandong Second Provincial General Hospital, Jinan, Shandong, China